CLINICAL TRIAL: NCT05415397
Title: Precision Psychiatry: Anti-inflammatory Medication in Immuno-metabolic Depression
Brief Title: Treating Immuno-metabolic Depression With Anti-inflammatory Drugs
Acronym: INFLAMED
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Netherlands Brain Foundation (Other)
Responsible Party: Principal Investigator, Yuri Milaneschi, Assistant Professor, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL79765.029.21
Record Dates: First submitted 2022-06-03; First posted 2022-06-13 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Depressive Disorder, Major; Inflammation
Keywords: INFLAMED; Depression; Inflammation; Immuno-metabolic Depression; Celecoxib
MeSH Terms: conditions — Depressive Disorder, Major; Inflammation; Depression | interventions — Celecoxib

STUDY DESIGN:
Intervention Model Description: 12-week double-blind, randomized (1:1), placebo-controlled trial comparing celecoxib add-on (400 mg/d) versus placebo add-on to TAU in the treatment of 140 subjects with MDD and Immuno-metabolic Depression features
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Celecoxib (Experimental): Celecoxib 400 mg/day, 2 capsules (200 mg) daily, 12 weeks
  Interventions: Drug: Celecoxib 400mg
- Placebo (Placebo Comparator): Placebo, 2 capsules daily, 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Celecoxib 400mg — Celecoxib add-on (400mg daily) add-on to treatment as usual (standard antidepressant treatment)
  Other Names: Celecoxib, ATC M01AH01
  Arms: Celecoxib
Drug: Placebo — Placebo add-on to treatment as usual (standard antidepressant treatment)
  Arms: Placebo

SUMMARY:
As the role of (neuro)inflammation in depression is emerging, augmentation of antidepressant treatments with anti-inflammatory drugs such as celecoxib has shown encouraging preliminary results. However, inflammation is not present in all depressed patients. Depression is heterogeneous: patients express diverse and sometimes opposing symptoms and biological profiles. The investigators of the present trial recently introduced the concept of ImmunoMetabolic Depression (IMD), characterized by the clustering of inflammatory/metabolic dysregulations and atypical, energy-related symptoms (hyperphagia, weight gain, hypersomnia, fatigue and leaden paralysis), and present in approximately 30% of cases. Converging evidence suggests that in this subgroup of depression cases, inflammation may exert a crucial pathobiological mechanism, representing therefore an actionable therapeutic target. In this trial IMD will be applied as a tool to personalize treatment, by matching depressed subjects with IMD with a targeted anti-inflammatory add-on treatment.

In this study, 140 persons with IMD will be selected. In this specific group of patients, the investigators will test whether celecoxib add-on (400 mg/d) is more effective than placebo in the treatment of depression through a 12-week double-blind, randomized (1:1), placebo-controlled trial. By selecting specifically depressed patients with IMD, the proposed treatment selectively targets key inflammatory pathophysiological pathways to enhance clinical outcome for depression. This personalized approach is expected to lead to large health gains for a sizable proportion of patients. The main hypothesis is that the group of patients with IMD receiving TAU + celecoxib, as compared to the TAU + placebo, will show a better symptom course over the 12-week follow-up.

DETAILED DESCRIPTION:
Rationale: Depression is a major driver of disability and related health-care costs. Available treatment options are far from optimal, with only ~60% response. Developing effective treatments requires new treatment targets to depression pathophysiology. As the role of (neuro)inflammation in depression is emerging, augmentation of antidepressant treatments with anti-inflammatory drugs such as celecoxib has shown encouraging preliminary results. However, inflammation is not present in all depressed patients. Depression is heterogeneous: patients express diverse and sometimes opposing symptoms and biological profiles. The investigators of the present study recently introduced the concept of ImmunoMetabolic Depression (IMD), characterized by the clustering of inflammatory/metabolic dysregulations and atypical, energy-related symptoms (hyperphagia, weight gain, hypersomnia, fatigue and leaden paralysis), and present in 30% of cases. Converging evidence suggests that in this subgroup of depression cases, inflammation may exert a crucial pathobiological mechanism, representing therefore an actionable therapeutic target. In this study IMD will be applied as a tool to personalize treatment, by matching depressed subjects with IMD with a targeted anti-inflammatory add-on treatment. The underlying hypothesis is that this personalized intervention in subjects with IMD, through a reduction of inflammation, lowers depressive symptoms and associated physical fatigue, while increasing functioning compared to placebo.

Objective: Among patients under treatment for depression, 140 persons with IMD will be selected. In this specific group of patients, the investigators will test whether celecoxib add-on (400 mg/d) is more effective than placebo in the treatment of depression through a 12-week double-blind, randomized (1:1), placebo-controlled trial.

Study design:12-week double-blind placebo-controlled randomized clinical trial Study population: 140 persons with major depressive disorder (DMS-5) with atypical, energy-related symptoms (≥6 on IDS atypical, energy-related symptoms) AND low-grade inflammation (CRP>1mg/L) (e.g. ImmunoMetabolic Depression), and under treatment with SSRI or SNRIs.

Intervention: celecoxib add-on (400 mg/d) vs placebo Main study parameters/endpoints: Primary outcome parameter is the difference in trajectories of depression symptoms, as measured with the 30-item Inventory of Depressive Symptomatology - self-report during follow-up. Secondary outcome parameters include amongst others, response on the IDS, remission, anxiety, fatigue, food craving, sleep and adverse side events.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of MDD confirmed with clinical interview (MINI-S voor DSM-5 Nederlandse versie 2019)
* Currently using pharmacotherapy (e.g., SSRI, SNRI, TCA, TetraCA, MAOI, other antidepressant [bupropion, vortioxetine, agomelatine])) and/or psychotherapy. Subjects should be on the current treatment for at least 4 weeks
* IDS-SR score ≥26 (moderate to severe depressive symptoms) and a score ≥6 on atypical, energy-related symptoms scale from IDS
* CRP > 1mg/L
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies: 1) is not a woman of child bearing potential (WOCBP); 2) Is a WOCBP and agrees to use, or is already using, a contraceptive method during the intervention period and up to 1 month after the intervention
* Signed informed consent

Exclusion Criteria:

* Contraindications for celecoxib (history of: peptic ulcers, gastrointestinal bleeding, ischemic heart disease, stroke, heart failure, allergic reactions to aspirin/NSAIDs/coxibs; impaired kidney function (creatinine clearance < 30 ml/min), impaired liver function (ALT > 2x ULT)
* ECT in the past 3 months
* Being on other psychotropic drugs
* Clinically overt alcohol/drug dependence or other primary psychiatric diagnoses (schizophrenia, schizoaffective, OCD, or bipolar disorder)
* Chronic use of anti-inflammatory drugs and corticosteroids
* Current use of anticoagulants
* Not speaking Dutch

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms severity | 12 weeks
  Depressive symptoms severity measured with the Inventory of Depressive Symptomatology - Self Report (IDS-SR; score ranging from 0 to 84, higher scores indicate higher severity of depressive symptoms). Trajectories of depressive symptoms will be modeled via mixed models including bi-weekly assessments

SECONDARY OUTCOMES:
Number of participants achieving Response | 12 weeks
  Response is defined as 50% reduction in depressive symptoms severity measured with Inventory of Depressive Symptomatology - Self Report (IDS-SR; score ranging from 0 to 84, higher scores indicate higher severity of depressive symptoms)
Number of participants achieving Remission | 12 weeks
  Remission is defined as absence of DSM-5 Major Depressive Disorder (MDD), identified using the Mini International Neuropsychiatric Interview - Simplified (MINI-S voor DSM-5 Nederlandse versie 2019)
Symptom profile: atypical, energy-related depressive symptoms (AES) | 12 weeks
  AES measured with 5 items (N 4, 12, 14, 20, 30) of the Inventory of Depressive Symptomatology - Self Report (IDS-SR). AES score ranging from 0 to 15, higher scores indicate higher severity of depressive symptoms.

OTHER OUTCOMES:
Fatigue | 12 weeks
  Fatigue measured by the Checklist Individuele Spankracht (CIS), which assess fatigue in 4 subscales: subjective experience of fatigue, reduction in motivation, reduction in activity and reduction in concentration. In each domain, higher scores indicate higher fatigue
Food craving | 12 weeks
  Food craving measured with General Food Craving Questionnaire Trait (G-FCQ-T; score ranging from 21 to 126, higher scores indicate more intense food craving)
Daytime sleepiness | 12 weeks
  Daytime sleepiness measured with the Epsworth Sleepiness Scale (ESS; score ranging from 0 to 24, higher scores indicates higher propensity to daytime sleepiness)
Night-time sleep | 12 weeks
  Sleep Duration measured with items 1,2,3 and 4 (self reports of bed time, asleep time, wake-time, sleep duration) of the Pittsburgh Sleep Quality Index (PSQI)
Anxiety symptoms | 12 weeks
  Anxiety symptoms measured with General Anxiety Disorder-7 (GAD-7, score ranging from 0 to 21, higher scores indicate higher anxiety)
Functionality | 12 weeks
  General functioning and disability measured with the WHO Disability Schedule (WHODAS, score ranging from 12 to 60, higher scores indicate more disability)
Pain severity | 12 weeks
  Pain measured by numeric rating scale (score ranging from 0 to 10, higher scores indicate higher pain)
Therapy compliance | 12 weeks
  Pill count
Inflammatory and metabolic blood markers | 12 weeks
  CRP, IL-6, TNF-α, cholesterol, triglycerides, glucose
Side effects | 12 weeks
  Side effects measured with the list applied in the PREDDICT RCT and theThe Antidepressant Side-Effect Checklist (ASEC-21)

CONTACTS AND LOCATIONS:
Overall Officials: Yuri Milaneschi, PhD, Principal Investigator — Amsterdam UMC, location VUmc; Femke Lamers, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- Department of Psychiatry Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Individual data collected during the study of participants explicitly agreeing on this possibility trough written informed consent; data will be de-identified
Supporting Information: Study Protocol
Time Frame: Immediately following study closure and publication of the main results, no end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose

REFERENCES:
- [Background] Milaneschi Y, Lamers F, Berk M, Penninx BWJH. Depression Heterogeneity and Its Biological Underpinnings: Toward Immunometabolic Depression. Biol Psychiatry. 2020 Sep 1;88(5):369-380. doi: 10.1016/j.biopsych.2020.01.014. Epub 2020 Jan 28. PMID 32247527
- [Background] Lamers F, Milaneschi Y, Vinkers CH, Schoevers RA, Giltay EJ, Penninx BWJH. Depression profilers and immuno-metabolic dysregulation: Longitudinal results from the NESDA study. Brain Behav Immun. 2020 Aug;88:174-183. doi: 10.1016/j.bbi.2020.04.002. Epub 2020 Apr 6. PMID 32272220
- [Background] Penninx BW, Milaneschi Y, Lamers F, Vogelzangs N. Understanding the somatic consequences of depression: biological mechanisms and the role of depression symptom profile. BMC Med. 2013 May 15;11:129. doi: 10.1186/1741-7015-11-129. PMID 23672628
- [Background] Milaneschi Y, Kappelmann N, Ye Z, Lamers F, Moser S, Jones PB, Burgess S, Penninx BWJH, Khandaker GM. Association of inflammation with depression and anxiety: evidence for symptom-specificity and potential causality from UK Biobank and NESDA cohorts. Mol Psychiatry. 2021 Dec;26(12):7393-7402. doi: 10.1038/s41380-021-01188-w. Epub 2021 Jun 16. PMID 34135474
- [Background] Kohler O, Benros ME, Nordentoft M, Farkouh ME, Iyengar RL, Mors O, Krogh J. Effect of anti-inflammatory treatment on depression, depressive symptoms, and adverse effects: a systematic review and meta-analysis of randomized clinical trials. JAMA Psychiatry. 2014 Dec 1;71(12):1381-91. doi: 10.1001/jamapsychiatry.2014.1611. PMID 25322082
- [Background] Kohler-Forsberg O, N Lydholm C, Hjorthoj C, Nordentoft M, Mors O, Benros ME. Efficacy of anti-inflammatory treatment on major depressive disorder or depressive symptoms: meta-analysis of clinical trials. Acta Psychiatr Scand. 2019 May;139(5):404-419. doi: 10.1111/acps.13016. Epub 2019 Mar 28. PMID 30834514
- [Background] Osimo EF, Baxter LJ, Lewis G, Jones PB, Khandaker GM. Prevalence of low-grade inflammation in depression: a systematic review and meta-analysis of CRP levels. Psychol Med. 2019 Sep;49(12):1958-1970. doi: 10.1017/S0033291719001454. Epub 2019 Jul 1. PMID 31258105
- [Background] Baune BT, Sampson E, Louise J, Hori H, Schubert KO, Clark SR, Mills NT, Fourrier C. No evidence for clinical efficacy of adjunctive celecoxib with vortioxetine in the treatment of depression: A 6-week double-blind placebo controlled randomized trial. Eur Neuropsychopharmacol. 2021 Dec;53:34-46. doi: 10.1016/j.euroneuro.2021.07.092. Epub 2021 Aug 8. PMID 34375789
- [Background] Strawbridge R, Arnone D, Danese A, Papadopoulos A, Herane Vives A, Cleare AJ. Inflammation and clinical response to treatment in depression: A meta-analysis. Eur Neuropsychopharmacol. 2015 Oct;25(10):1532-43. doi: 10.1016/j.euroneuro.2015.06.007. Epub 2015 Jun 20. PMID 26169573
- [Derived] Zwiep JC, Bet PM, Rhebergen D, Nurmohamed MT, Vinkers CH, Penninx BWJH, Milaneschi Y, Lamers F. Efficacy of celecoxib add-on treatment for immuno-metabolic depression: Protocol of the INFLAMED double-blind placebo-controlled randomized controlled trial. Brain Behav Immun Health. 2022 Dec 30;27:100585. doi: 10.1016/j.bbih.2022.100585. eCollection 2023 Feb. PMID 36655056
- See also: Study website — https://immunometaboledepressie.nl/